CLINICAL TRIAL: NCT00538850
Title: A Randomized, Double-blind, Placebo-controlled Multi-center Study to Evaluate the Safety and Efficacy of Fentanyl Sublingual Spray (Fentanyl SL Spray) for the Treatment of Breakthrough Cancer Pain
Brief Title: Fentanyl Sublingual Spray in Treating Patients With Breakthrough Cancer Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: INS-05-001; CDR0000581128 (Registry Identifier: PDQ (Physician Data Query)); NCT00589342 (obsolete NCT alias)
Record Dates: First submitted 2007-10-01; First posted 2007-10-03 (Estimated); Results first posted 2014-03-05 (Estimated); Last update posted 2014-03-05 (Estimated); Status verified 2014-01

CONDITIONS: Cancer
Keywords: unspecified adult solid tumor, protocol specific; pain; adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with t(15;17)(q22;q12); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with t(8;21)(q22;q22); stage IV chronic lymphocytic leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic myelomonocytic leukemia; chronic phase chronic myelogenous leukemia; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III adult Burkitt lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III adult lymphoblastic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage III mantle cell lymphoma; stage IV adult Burkitt lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV adult lymphoblastic lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma; stage IV mantle cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent small lymphocytic lymphoma; recurrent marginal zone lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; recurrent mycosis fungoides/Sezary syndrome; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma; de novo myelodysplastic syndromes; myelodysplastic/myeloproliferative neoplasm, unclassifiable; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; atypical chronic myeloid leukemia, BCR-ABL1 negative; stage II adult Hodgkin lymphoma; stage III adult Hodgkin lymphoma; stage IV adult Hodgkin lymphoma; contiguous stage II adult Burkitt lymphoma; stage I adult Burkitt lymphoma; contiguous stage II adult diffuse large cell lymphoma; contiguous stage II adult diffuse mixed cell lymphoma; contiguous stage II adult diffuse small cleaved cell lymphoma; contiguous stage II small lymphocytic lymphoma; contiguous stage II marginal zone lymphoma; stage I adult diffuse large cell lymphoma; stage I adult diffuse mixed cell lymphoma; stage I adult diffuse small cleaved cell lymphoma; stage I small lymphocytic lymphoma; stage I marginal zone lymphoma; contiguous stage II grade 1 follicular lymphoma; contiguous stage II grade 2 follicular lymphoma; contiguous stage II grade 3 follicular lymphoma; stage I grade 1 follicular lymphoma; stage I grade 2 follicular lymphoma; stage I grade 3 follicular lymphoma; contiguous stage II mantle cell lymphoma; stage I mantle cell lymphoma; contiguous stage II adult immunoblastic large cell lymphoma; stage I adult immunoblastic large cell lymphoma; contiguous stage II adult lymphoblastic lymphoma; stage I adult lymphoblastic lymphoma; refractory multiple myeloma; anaplastic large cell lymphoma; angioimmunoblastic T-cell lymphoma; recurrent adult T-cell leukemia/lymphoma; stage I adult T-cell leukemia/lymphoma; stage II adult T-cell leukemia/lymphoma; stage III adult T-cell leukemia/lymphoma; stage IV adult T-cell leukemia/lymphoma; stage I cutaneous T-cell non-Hodgkin lymphoma; stage II cutaneous T-cell non-Hodgkin lymphoma; stage III cutaneous T-cell non-Hodgkin lymphoma; stage IV cutaneous T-cell non-Hodgkin lymphoma; stage I mycosis fungoides/Sezary syndrome; stage II mycosis fungoides/Sezary syndrome; stage III mycosis fungoides/Sezary syndrome; stage IV mycosis fungoides/Sezary syndrome; chronic eosinophilic leukemia; primary myelofibrosis; chronic neutrophilic leukemia; essential thrombocythemia; polycythemia vera; relapsing chronic myelogenous leukemia; T-cell large granular lymphocyte leukemia; recurrent adult acute lymphoblastic leukemia; recurrent adult acute myeloid leukemia; untreated adult acute lymphoblastic leukemia; untreated adult acute myeloid leukemia; secondary acute myeloid leukemia; acute undifferentiated leukemia; refractory chronic lymphocytic leukemia; stage 0 chronic lymphocytic leukemia; stage I chronic lymphocytic leukemia; stage II chronic lymphocytic leukemia; stage III chronic lymphocytic leukemia; refractory hairy cell leukemia; progressive hairy cell leukemia, initial treatment; prolymphocytic leukemia; recurrent adult grade III lymphomatoid granulomatosis; Waldenström macroglobulinemia; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; post-transplant lymphoproliferative disorder; extramedullary plasmacytoma; isolated plasmacytoma of bone; monoclonal gammopathy of undetermined significance; primary systemic amyloidosis; adult acute lymphoblastic leukemia in remission; adult acute myeloid leukemia in remission; adult grade III lymphomatoid granulomatosis; AIDS-related peripheral/systemic lymphoma; AIDS-related primary CNS lymphoma; intraocular lymphoma; meningeal chronic myelogenous leukemia; primary central nervous system non-Hodgkin lymphoma; primary central nervous system Hodgkin lymphoma; stage I adult Hodgkin lymphoma; recurrent squamous cell carcinoma of the hypopharynx; stage I squamous cell carcinoma of the hypopharynx; stage II squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage I squamous cell carcinoma of the larynx; stage I verrucous carcinoma of the larynx; stage II squamous cell carcinoma of the larynx; stage II verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage I adenoid cystic carcinoma of the oral cavity; stage I mucoepidermoid carcinoma of the oral cavity; stage I verrucous carcinoma of the oral cavity; stage II adenoid cystic carcinoma of the oral cavity; stage II mucoepidermoid carcinoma of the oral cavity; stage II verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; stage I squamous cell carcinoma of the lip and oral cavity; stage II squamous cell carcinoma of the lip and oral cavity; stage III squamous cell carcinoma of the lip and oral cavity; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage I basal cell carcinoma of the lip; stage II basal cell carcinoma of the lip; stage III basal cell carcinoma of the lip; stage IV basal cell carcinoma of the lip; metastatic squamous neck cancer with occult primary squamous cell carcinoma; recurrent metastatic squamous neck cancer with occult primary; untreated metastatic squamous neck cancer with occult primary; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage I lymphoepithelioma of the nasopharynx; stage I squamous cell carcinoma of the nasopharynx; stage II lymphoepithelioma of the nasopharynx; stage II squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage I lymphoepithelioma of the oropharynx; stage I squamous cell carcinoma of the oropharynx; stage II lymphoepithelioma of the oropharynx; stage II squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage I esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage I inverted papilloma of the paranasal sinus and nasal cavity; stage I midline lethal granuloma of the paranasal sinus and nasal cavity; stage I squamous cell carcinoma of the paranasal sinus and nasal cavity; stage II esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage II inverted papilloma of the paranasal sinus and nasal cavity; stage II midline lethal granuloma of the paranasal sinus and nasal cavity; stage II squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; high-grade salivary gland mucoepidermoid carcinoma; low-grade salivary gland mucoepidermoid carcinoma; recurrent salivary gland cancer; salivary gland acinic cell tumor; salivary gland adenocarcinoma; salivary gland adenoid cystic carcinoma; salivary gland anaplastic carcinoma; salivary gland malignant mixed cell type tumor; salivary gland poorly differentiated carcinoma; salivary gland squamous cell carcinoma; stage I salivary gland cancer; stage II salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; adult grade I meningioma; adult choroid plexus tumor; adult craniopharyngioma; adult myxopapillary ependymoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult pineocytoma; adult ependymoma; adult subependymoma; adult oligodendroglioma; adult subependymal giant cell astrocytoma; meningeal melanocytoma; adult meningeal hemangiopericytoma; adult pineal gland astrocytoma; adult central nervous system germ cell tumor; adult medulloblastoma; adult supratentorial primitive neuroectodermal tumor (PNET); adult ependymoblastoma; adult anaplastic astrocytoma; adult anaplastic ependymoma; adult glioblastoma; adult gliosarcoma; adult giant cell glioblastoma; adult grade III meningioma; adult anaplastic oligodendroglioma; adult pineoblastoma; adult mixed glioma; recurrent adult brain tumor; adult anaplastic meningioma; adult papillary meningioma; adult brain stem glioma; stage IA cervical cancer; stage IB cervical cancer; stage IIA cervical cancer; stage IIB cervical cancer; stage III cervical cancer; stage IVA cervical cancer; stage IVB cervical cancer; recurrent cervical cancer; recurrent endometrial carcinoma; stage I endometrial carcinoma; stage II endometrial carcinoma; stage III endometrial carcinoma; stage IV endometrial carcinoma; fallopian tube cancer; recurrent ovarian epithelial cancer; recurrent ovarian germ cell tumor; stage I ovarian epithelial cancer; stage I ovarian germ cell tumor; stage II ovarian epithelial cancer; stage II ovarian germ cell tumor; stage III ovarian epithelial cancer; stage III ovarian germ cell tumor; stage IV ovarian epithelial cancer; stage IV ovarian germ cell tumor; ovarian sarcoma; ovarian stromal cancer; recurrent uterine sarcoma; stage I uterine sarcoma; stage II uterine sarcoma; stage III uterine sarcoma; stage IV uterine sarcoma; recurrent colon cancer; stage I colon cancer; stage II colon cancer; stage III colon cancer; stage IV colon cancer; recurrent bladder cancer; recurrent gallbladder cancer; stage I bladder cancer; stage II bladder cancer; stage III bladder cancer; stage IV bladder cancer; recurrent gastric cancer; stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; advanced adult primary liver cancer; recurrent small intestine cancer; localized transitional cell cancer of the renal pelvis and ureter; metastatic transitional cell cancer of the renal pelvis and ureter; recurrent renal cell cancer; recurrent transitional cell cancer of the renal pelvis and ureter; regional transitional cell cancer of the renal pelvis and ureter; stage I renal cell cancer; stage II renal cell cancer; stage III renal cell cancer; stage IV renal cell cancer; distal urethral cancer; proximal urethral cancer; recurrent urethral cancer; urethral cancer associated with invasive bladder cancer; stage I adrenocortical carcinoma; stage II adrenocortical carcinoma; stage III adrenocortical carcinoma; stage IV adrenocortical carcinoma; recurrent adrenocortical carcinoma; extragonadal germ cell tumor; localized gastrointestinal carcinoid tumor; metastatic gastrointestinal carcinoid tumor; recurrent gastrointestinal carcinoid tumor; regional gastrointestinal carcinoid tumor; gastrinoma; insulinoma; WDHA syndrome; glucagonoma; pancreatic polypeptide tumor; somatostatinoma; recurrent islet cell carcinoma; carcinoma of the appendix; localized extrahepatic bile duct cancer; recurrent extrahepatic bile duct cancer; unresectable extrahepatic bile duct cancer; localized gallbladder cancer; unresectable gallbladder cancer; gastrointestinal stromal tumor; localized resectable adult primary liver cancer; localized unresectable adult primary liver cancer; recurrent adult primary liver cancer; stage I pancreatic cancer; stage II pancreatic cancer; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer; small intestine adenocarcinoma; small intestine leiomyosarcoma; small intestine lymphoma; stage I non-small cell lung cancer; stage II non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; recurrent non-small cell lung cancer; pulmonary carcinoid tumor; extensive stage small cell lung cancer; limited stage small cell lung cancer; recurrent small cell lung cancer; liver metastases; lung metastases; primary peritoneal cavity cancer; lung papilloma; peripheral primitive neuroectodermal tumor of the kidney; clear cell sarcoma of the kidney; rhabdoid tumor of the kidney; congenital mesoblastic nephroma; stage II breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; recurrent breast cancer; male breast cancer; breast cancer in situ; localized osteosarcoma; metastatic osteosarcoma; recurrent osteosarcoma; localized Ewing sarcoma/peripheral primitive neuroectodermal tumor; metastatic Ewing sarcoma/peripheral primitive neuroectodermal tumor; recurrent Ewing sarcoma/peripheral primitive neuroectodermal tumor; chondrosarcoma; malignant giant cell tumor of bone; desmoid tumor; stage I adult soft tissue sarcoma; stage II adult soft tissue sarcoma; stage III adult soft tissue sarcoma; stage IV adult soft tissue sarcoma; recurrent adult soft tissue sarcoma; recurrent thymoma and thymic carcinoma; advanced malignant mesothelioma; localized malignant mesothelioma; recurrent malignant mesothelioma; phosphaturic mesenchymal tumor; stage I malignant testicular germ cell tumor; stage II malignant testicular germ cell tumor; stage III malignant testicular germ cell tumor; recurrent malignant testicular germ cell tumor; stage 0 penile cancer; stage I penile cancer; stage II penile cancer; stage III penile cancer; stage IV penile cancer; recurrent penile cancer; stage I prostate cancer; stage IIB prostate cancer; stage IIA prostate cancer; stage III prostate cancer; stage IV prostate cancer; recurrent prostate cancer; stage 0 vaginal cancer; stage I vaginal cancer; stage II vaginal cancer; stage III vaginal cancer; stage IVA vaginal cancer; stage IVB vaginal cancer; recurrent vaginal cancer; stage 0 vulvar cancer; stage I vulvar cancer; stage II vulvar cancer; stage III vulvar cancer; stage IVB vulvar cancer; recurrent vulvar cancer; stage 0 anal cancer; stage I anal cancer; stage II anal cancer; stage IIIA anal cancer; stage IIIB anal cancer; stage IV anal cancer; recurrent anal cancer; stage 0 rectal cancer; stage I rectal cancer; stage II rectal cancer; stage III rectal cancer; stage IV rectal cancer; recurrent rectal cancer; stage 0 esophageal cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; stage I thymoma; stage II thymoma; stage III thymoma; stage IVA thymoma; stage IVB thymoma; recurrent melanoma; stage 0 melanoma; stage IA melanoma; stage IB melanoma; stage IIA melanoma; stage IIB melanoma; stage IIC melanoma; stage IIIA melanoma; stage IIIB melanoma; stage IIIC melanoma; stage IV melanoma
MeSH Terms: conditions — Neoplasms; Pain; Congenital Abnormalities; Leukemia, Lymphocytic, Chronic, B-Cell; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Chronic-Phase; Burkitt Lymphoma; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, B-Cell, Marginal Zone; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Hodgkin Disease; Lymphoma, T-Cell, Cutaneous; Mycosis Fungoides; Sezary Syndrome; Multiple Myeloma; Myeloproliferative Disorders; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Lymphoma, Large-Cell, Anaplastic; Immunoblastic Lymphadenopathy; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma; Pdgfra-Associated Chronic Eosinophilic Leukemia; Primary Myelofibrosis; Leukemia, Neutrophilic, Chronic; Thrombocythemia, Essential; Polycythemia Vera; Leukemia, Large Granular Lymphocytic; Leukemia, Myeloid, Acute; Leukemia, Biphenotypic, Acute; Leukemia, Hairy Cell; Leukemia, Prolymphocytic; Waldenstrom Macroglobulinemia; Monoclonal Gammopathy of Undetermined Significance; Immunoglobulin Light-chain Amyloidosis; Intraocular Lymphoma; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Choroid Plexus Neoplasms; Craniopharyngioma; Ependymoma; Astrocytoma; Pinealoma; Glioma, Subependymal; Oligodendroglioma; Medulloblastoma; Neuroectodermal Tumors, Primitive; Glioblastoma; Gliosarcoma; Meningioma; Glioma; Brain Neoplasms; Uterine Cervical Neoplasms; Endometrial Neoplasms; Fallopian Tube Neoplasms; Carcinoma, Ovarian Epithelial; Colonic Neoplasms; Urinary Bladder Neoplasms; Gallbladder Neoplasms; Stomach Neoplasms; Carcinoma, Renal Cell; Urethral Neoplasms; Adrenocortical Carcinoma; Gastrinoma; Insulinoma; Vipoma; Glucagonoma; Somatostatinoma; Carcinoma, Islet Cell; Appendiceal Neoplasms; Bile Duct Neoplasms; Gastrointestinal Stromal Tumors; Carcinoma, Hepatocellular; Pancreatic Neoplasms; Carcinoma, Non-Small-Cell Lung; Small Cell Lung Carcinoma; Nephroma, Mesoblastic; Breast Neoplasms; Breast Neoplasms, Male; Breast Carcinoma In Situ; Osteosarcoma; Neuroectodermal Tumors, Primitive, Peripheral; Chondrosarcoma; Desmoid Tumors; Sarcoma; Thymoma; Mesothelioma, Malignant; Testicular Neoplasms; Penile Neoplasms; Prostatic Neoplasms; Vaginal Neoplasms; Vulvar Neoplasms; Anus Neoplasms; Rectal Neoplasms; Esophageal Neoplasms; Melanoma | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- Fentanyl sublingual spray (Experimental): Participants received fentanyl sublingual spray 7 times or placebo 3 times in random order to treat up to a maximum of 2 breakthrough pain episodes per day with a minimum separation of 2 hours between treatments. Patients received a dose of 100 to 1600 µg determined in the open-label dose titration period of the current study.
  Interventions: Drug: Fentanyl sublingual spray; Drug: Placebo

INTERVENTIONS:
Drug: Fentanyl sublingual spray — In the open-label titration period of the study, participants started at a dose of 100, 200, or 400 µg and titrated upward to a maximum dose of 1600 µg. Titration was stopped when the dose administered provided adequate analgesia for breakthrough pain without unacceptable side effects or the maximum titration period of 21±5 days was reached. In the double-blind period of the study, participants received fentanyl sublingual spray in doses of 100, 200, 400, 600, 800, 1200, or 1600 µg determined in the open-label titration period of the study.
  Other Names: SUBSYS
Drug: Placebo — Matching placebo to fentanyl sublingual spray.

SUMMARY:
This is a phase III, randomized, double-blind, placebo-controlled, multicenter study of the clinical response to fentanyl sublingual spray as a treatment for breakthrough cancer pain. The study medication is administered under the tongue as a simple spray and can be self-administered by patients or assisted by their caregivers. Patients are titrated to an effective-dose of fentanyl sublingual spray in the open-label titration period and then proceed to the double-blind randomized period where they randomly receive 7 treatments with fentanyl sublingual spray and 3 treatments with placebo. Patients are treated for up to a total of 6-7 weeks (including both the open-label titration and the double-blind randomized periods).

DETAILED DESCRIPTION:
RATIONALE

Fentanyl sublingual spray may help relieve breakthrough pain in patients receiving opioids for cancer pain.

OBJECTIVES

Primary

* Determine the efficacy and safety of fentanyl sublingual spray for the treatment of breakthrough cancer pain in patients on around-the-clock opioids for their persistent cancer pain.

Secondary

* Evaluate the safety of fentanyl sublingual spray in these opioid-tolerant patients.
* Assess the patient's satisfaction with treatment medication.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥ 18 years of age.
* Diagnosis of cancer.
* Opioid-tolerant. Subjects who were opioid tolerant were those taking ≥ 60 mg of oral morphine/day, at least 25 μg of transdermal fentanyl/hour, at least 30 mg of oxycodone daily, at least 8 mg of oral hydromorphone daily or an equianalgesic dose of another opioid for a week or longer for cancer-related pain.
* Experienced persistent pain related to the cancer or its treatment of moderate or lesser intensity in the 24 hours prior to assessment by a verbal rating scale at the Screening Visit.
* Over the previous 7 days, subject experienced, on average, 1 to 4 breakthrough cancer pain episodes per day usually at least partially controlled by supplemental medication of at least 5 mg immediate-release morphine or an equivalent short-acting opioid (eg, oxycodone, hydrocodone, or codeine with acetaminophen).
* Able to evaluate and record pain relief, assess medication performance at set times after dosing, record AEs, record each use of the study drug or supplemental medication in an electronic diary (a caregiver may have provided the subject the medication, help with the mechanics of handling the electronic diary but was not permitted to record any information in the electronic diary).
* Able and willing to give informed consent.
* Women of childbearing potential were to have a) a negative serum pregnancy test, b) not be breastfeeding and c) agree to practice a reliable form of contraception.

Exclusion Criteria:

* Intolerance to opioids or fentanyl.
* Current use of commercially available oral short-acting fentanyl for breakthrough pain. Subjects previously on Actiq or Fentora were permitted to be enrolled if they had a 7 day washout.
* Rapidly increasing/uncontrolled pain.
* A history of major organ system impairment or disease, that in the Investigator's or his/her designee's opinion could increase the risk associated with the use of opioids.
* Uncontrolled hypertension (systolic blood pressure {SBP} > 180 mmHg or diastolic blood pressure [DBP] > 90 mmHg on 2 occasions ≥ 6 hours apart) despite antihypertensive therapy, or a history of hypertensive crisis within the past 2 years.
* A recent history (≤ 2 years prior) of transient ischemic attacks, neural vascular disease, stroke, or cerebral aneurysms.
* Clinically uncontrolled sleep apnea.
* Brain metastases with signs or symptoms of increased intracranial pressure.
* Inability to assess pain or response to pain medications for any reason, including psychiatric disorder, concurrent medical disorder, or concomitant therapy.
* Received investigational study product(s) ≤ 30 days prior to the Screening Visit.
* Painful erythema, oedema or ulcers under the tongue.
* Use of monoamine oxidase (MAO) inhibitors within 14 days of the Screening Visit.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2007-10; Primary Completion 2010-02 (Actual); Study Completion 2010-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Larry Dillaha, MD, Study Chair — INSYS Therapeutics Inc
Locations (1):
- InSys Therapeutics, Incorporated, Chandler, Arizona, United States

REFERENCES:
- [Result] Rauck R, Reynolds L, Geach J, Bull J, Stearns L, Scherlis M, Parikh N, Dillaha L. Efficacy and safety of fentanyl sublingual spray for the treatment of breakthrough cancer pain: a randomized, double-blind, placebo-controlled study. Curr Med Res Opin. 2012 May;28(5):859-70. doi: 10.1185/03007995.2012.683111. Epub 2012 May 2. PMID 22480131
- [Derived] Alberts DS, Smith CC, Parikh N, Rauck RL. Fentanyl sublingual spray for breakthrough cancer pain in patients receiving transdermal fentanyl. Pain Manag. 2016 Oct;6(5):427-34. doi: 10.2217/pmt-2015-0009. Epub 2016 Mar 29. PMID 27020837

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: As there are dozens, if not hundreds, of cross-over sequences during the double-blind period of this study, instead of reporting participant flow for each of the cross-over sequences, participant flow is reported separately for the fentanyl and placebo groups.
Groups:
- Fentanyl Sublingual Spray - Titration: In the open-label titration period of the study, participants started at a dose of 100, 200, or 400 µg and titrated upward to a maximum dose of 1600 µg. Titration was stopped when the dose administered provided adequate analgesia for breakthrough pain without unacceptable side effects or the maximum titration period of 21±5 days was reached.
- Fentanyl Sublingual Spray - Double-blind: Participants received fentanyl sublingual spray 7 times randomly (out of 10 treatments total) to treat up to a maximum of 2 breakthrough pain episodes per day with a minimum separation of 2 hours between treatments. Patients received a dose of 100 to 1600 µg determined in the open-label dose titration period of the current study.
- Placebo - Double-blind: Participants received placebo 3 times randomly (out of 10 treatments total) to treat up to a maximum of 2 breakthrough pain episodes per day with a minimum separation of 2 hours between treatments. Patients received a dose of 100 to 1600 µg determined in the open-label dose titration period of the current study.
Period: Titration Period
Arm/Group | Fentanyl Sublingual Spray - Titration | Fentanyl Sublingual Spray - Double-blind | Placebo - Double-blind
Started | 130 | 0 (There were no participants in this reporting group in the titration period.) | 0 (There were no participants in this reporting group in the titration period.)
Completed | 98 | 0 | 0
Not Completed | 32 | 0 | 0
Period: Fentanyl Sublingual Spray - Double-blind
Arm/Group | Fentanyl Sublingual Spray - Titration | Fentanyl Sublingual Spray - Double-blind | Placebo - Double-blind
Started | 0 (There were no participants in this reporting group in the double-blind period.) | 98 | 0 (There were no participants in this reporting group in the double-blind period.)
Completed | 0 | 95 | 0
Not Completed | 0 | 3 | 0
Period: Placebo - Double-blind
Arm/Group | Fentanyl Sublingual Spray - Titration | Fentanyl Sublingual Spray - Double-blind | Placebo - Double-blind
Started | 0 (There were no participants in this reporting group in the double-blind period.) | 0 (There were no participants in this reporting group in the double-blind period.) | 98
Completed | 0 | 0 | 95
Not Completed | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Arm/Group | Fentanyl Sublingual Spray
Number analyzed (Participants) | 130
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.6 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 69
  Male | 61

OUTCOME MEASURES:

1. Primary Outcome: Summed Pain Intensity Differences (SPID) at 30 Minutes After Dosing (SPID30)
Description: Pain intensity was assessed by the participant using a 0-100 mm visual analog scale where 0 represented "no pain" and 100 represented "worst possible pain" at 0 (baseline, beginning of the pain episode), 5, 10, 15, and 30 minutes after each dose of study medication during each breakthrough pain episode. The pain intensity difference was defined as the difference in pain intensity at the various time points versus time 0 (baseline). SPID30 was calculated as the time-weighted sum of the PID scores using the following formula: SPID30=(5*PID5)+(5*PID10)+(5*PID15)+(15*PID30). The minimum and maximum SPID30 scores were -3000 and 3000. A higher score indicates less pain.
Time Frame: Baseline (time 0, beginning of each pain episode) through 30 minutes after dosing for each pain episode
Population: Intent-to-treat (ITT) population: All participants in the double-blind treatment period who received at least 1 dose of study medication and had at least 1 pain measurement. 4 of the 96 participants in the ITT population were excluded from analysis because they did not have at least 1 dose of study medication and 1 dose of placebo.
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Fentanyl Sublingual Spray: Participants received fentanyl sublingual spray 7 times randomly (out of 10 treatments total) to treat up to a maximum of 2 breakthrough pain episodes per day with a minimum separation of 2 hours between treatments. Patients received a dose of 100 to 1600 µg determined in the open-label dose titration period of the current study.
- Placebo: Participants received placebo 3 times randomly (out of 10 treatments total) to treat up to a maximum of 2 breakthrough pain episodes per day with a minimum separation of 2 hours between treatments. Patients received a dose of 100 to 1600 µg determined in the open-label dose titration period of the current study.
Arm/Group | Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 92 | 92
Units on a scale | 640.3 (458.8) | 399.6 (391.2)

2. Secondary Outcome: Summed Pain Intensity Differences (SPID) at 5, 10, 15, 45, and 60 Minutes After Dosing
Description: Pain intensity was assessed by the participant using a 0-100 mm visual analog scale where 0 represented "no pain" and 100 represented "worst possible pain" at 0 (baseline, beginning of the pain episode), 5, 10, 15, 30, 45 and 60 minutes after each dose of study medication during each breakthrough pain episode. The pain intensity difference was defined as the difference in pain intensity at the various time points versus time 0 (baseline). SPID was calculated as the time-weighted sum of the PID scores using the following formulas: SPID5=(5*PID5), SPID10=(5*PID5)+(5*PID10), SPID15=(5*PID5)+(5*PID10)+(5*PID15), SPID30=(5*PID5)+(5*PID10)+(5*PID15)+(15*PID30), SPID45=(5*PID5)+(5*PID10)+(5*PID15)+(15*PID30)+(15*PID45), SPID60=(5*PID5)+(5*PID10)+(5*PID15)+(15*PID30) +(15*PID45) +(15*PID60). The minimum and maximum SPID scores were -500 to 500, -1000 to 1000, -1500 to 1500, -3000 to 3000, -4500 to 4500, and -6000 to 6000, respectively. A higher score indicates less pain.
Time Frame: Baseline (time 0, beginning of each pain episode) through 60 minutes after dosing for each pain episode
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 92 | 92
Units on a scale
  SPID5 | 40.3 (57.7) | 32.0 (52.1)
  SPID10 | 115.0 (130.7) | 81.1 (108.0)
  SPID15 | 220.6 (209.7) | 150.3 (172.5)
  SPID45 | 1122.0 (731.9) | 667.0 (614.5)
  SPID60 | 1649.0 (1016.2) | 965.7 (862.1)

3. Secondary Outcome: Total Pain Relief (TOTPAR) at 5, 10, 15, 30, 45, and 60 Minutes After Dosing
Description: Pain relief (PAR) was assessed by the participant on a 5-point scale (1=No relief, 2=A little relief, 3=Moderate relief, 4=A lot of relief, 5=Complete relief) at 5, 10, 15, 30, 45 and 60 minutes after each dose of study medication during each breakthrough pain episode. TOTPAR was calculated as the time-weighted sum of the PAR scores at each time point using the following formulas: TOTPAR5=(5*PAR5), TOTPAR10=(5*PAR5)+(5*PAR10), TOTPAR15=(5*PAR5)+(5*PAR10)+(5*PAR15), TOTPAR30=(5*PAR5)+(5*PAR10)+(5*PAR15)+(15*PAR30), TOTPAR45=(5*PAR5)+(5*PAR10)+(5*PAR15)+(15*PAR30)+(15*PAR45), TOTPAR60=(5*PAR5)+(5*PAR10)+(5*PAR15)+(15*PAR30) +(15*PAR45) +(15*PAR60). The minimum and maximum TOTPAR5, TOTPAR10, TOTPAR15, TOTPAR30, TOTPAR45, and TOTPAR60 scores were 5 to 25, 10 to 50, 15 to 75, 30 to 150, 45 to 225, and 60 to 300, respectively. A higher score indicates more pain relief.
Time Frame: 5 through 60 minutes after dosing for each pain episode
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 92 | 92
Units on a scale
  TOTPAR5 | 8.6 (3.5) | 7.6 (3.3)
  TOTPAR10 | 19.7 (7.0) | 16.7 (6.5)
  TOTPAR15 | 32.9 (10.3) | 27.1 (10.0)
  TOTPAR30 | 78.3 (20.4) | 61.0 (20.8)
  TOTPAR45 | 126.3 (30.9) | 95.5 (32.0)
  TOTPAR60 | 176.4 (41.5) | 131.2 (43.6)

4. Secondary Outcome: Global Evaluation of the Study Medication at 30 and 60 Minutes After Dosing
Description: Global evaluation of the study medication was assessed by the participant on a 5-point scale (1=Poor, 2=Fair, 3=Good, 4=Very good, 5=Excellent) at 30 and 60 minutes after each dose of study medication during each breakthrough pain episode. A higher score indicates a better evaluation.
Time Frame: 30 through 60 minutes after dosing for each pain episode
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Fentanyl Sublingual Spray | Placebo
Number analyzed (Participants) | 92 | 92
Units on a scale
  30 minutes | 2.8 (0.8) | 2.0 (0.8)
  60 minutes | 3.1 (0.8) | 2.2 (0.8)

ADVERSE EVENTS:
Time Frame: All adverse events were followed to resolution, an outcome was reached, stabilization, or the event was otherwise explained regardless of whether the subject was still participating in the study.
Description: Safety population: All enrolled subjects who took at least 1 dose of fentanyl sublingual spray.
  As subjects may have taken both treatments on the same day and adverse events were only collected once each day, it is not possible to report adverse events separately for the 2 treatments.
Groups:
- Fentanyl Sublingual Spray - Double-blind: Participants received fentanyl sublingual spray 7 times or placebo 3 times in random order to treat up to a maximum of 2 breakthrough pain episodes per day with a minimum separation of 2 hours between treatments. Patients received a dose of 100 to 1600 µg determined in the open-label dose titration period of the current study.
Arm/Group | Fentanyl Sublingual Spray - Titration | Fentanyl Sublingual Spray - Double-blind
Serious Adverse Events (participants affected / at risk) | 7/130 | 6/98
Other Adverse Events (participants affected / at risk) | 78/130 | 47/98
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fentanyl Sublingual Spray - Titration (N=130) | Fentanyl Sublingual Spray - Double-blind (N=98)
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 1 | 1
Vomiting (Gastrointestinal disorders) | 1 | 1
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 1 | 0
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Tachycardia (Cardiac disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Fentanyl Sublingual Spray - Titration (N=130) | Fentanyl Sublingual Spray - Double-blind (N=98)
Nausea (Gastrointestinal disorders) | 17 | 7
Vomiting (Gastrointestinal disorders) | 10 | 4
Diarrhoea (Gastrointestinal disorders) | 7 | 3
Constipation (Gastrointestinal disorders) | 5 | 0
Stomatitis (Gastrointestinal disorders) | 5 | 1
Dry mouth (Gastrointestinal disorders) | 2 | 2
Abdominal discomfort (Gastrointestinal disorders) | 1 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 1 | 0
Flatulence (Gastrointestinal disorders) | 1 | 1
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastrointestinal motility disorder (Gastrointestinal disorders) | 1 | 0
Gingival hyperplasia (Gastrointestinal disorders) | 1 | 0
Glossitis (Gastrointestinal disorders) | 1 | 0
Hyperchlorhydria (Gastrointestinal disorders) | 1 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 1 | 0
Odynophagia (Gastrointestinal disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 1 | 0
Retching (Gastrointestinal disorders) | 1 | 1
Tongue ulceration (Gastrointestinal disorders) | 1 | 0
Somnolence (Nervous system disorders) | 11 | 2
Dizziness (Nervous system disorders) | 10 | 2
Headache (Nervous system disorders) | 5 | 3
Sedation (Nervous system disorders) | 4 | 0
Dysgeusia (Nervous system disorders) | 3 | 0
Lethargy (Nervous system disorders) | 2 | 0
Areflexia (Nervous system disorders) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Burning sensation (Nervous system disorders) | 1 | 0
Disturbance In attention (Nervous system disorders) | 1 | 0
Dyskinesia (Nervous system disorders) | 1 | 0
Facial palsy (Nervous system disorders) | 1 | 0
Hyperreflexia (Nervous system disorders) | 1 | 0
Hypoaesthesia (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Pyrexia (General disorders) | 8 | 1
Oedema peripheral (General disorders) | 7 | 5
Asthenia (General disorders) | 4 | 2
Fatigue (General disorders) | 4 | 2
Application site irritation (General disorders) | 3 | 0
Adverse drug reaction (General disorders) | 1 | 0
Catheter related complication (General disorders) | 1 | 0
Catheter site erythema (General disorders) | 1 | 0
Chest discomfort (General disorders) | 1 | 1
Feeling abnormal (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 1 | 0
Pain (General disorders) | 1 | 1
Thirst (General disorders) | 1 | 0
Urinary tract infection (Infections and infestations) | 5 | 3
Cellulitis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 1
Oral herpes (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 1 | 1
Pyelonephritis (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Increased bronchial secretion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Confusional state (Psychiatric disorders) | 4 | 0
Insomnia (Psychiatric disorders) | 4 | 1
Agitation (Psychiatric disorders) | 2 | 0
Hallucination (Psychiatric disorders) | 2 | 0
Anxiety (Psychiatric disorders) | 1 | 1
Depression (Psychiatric disorders) | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0
Mood swings (Psychiatric disorders) | 1 | 0
Paranoia (Psychiatric disorders) | 1 | 0
Restlessness (Psychiatric disorders) | 1 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 2 | 5
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 0
Blister (Skin and subcutaneous tissue disorders) | 1 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Skin lesion (Skin and subcutaneous tissue disorders) | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 2 | 0
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1 | 0
Mobility decreased (Musculoskeletal and connective tissue disorders) | 1 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0
Anorexia (Metabolism and nutrition disorders) | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Decreased appetite (Metabolism and nutrition disorders) | 1 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0
Increased appetite (Metabolism and nutrition disorders) | 1 | 0
Malnutrition (Metabolism and nutrition disorders) | 1 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Spinal cord neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Urinary retention (Renal and urinary disorders) | 3 | 0
Bladder distension (Renal and urinary disorders) | 1 | 0
Bladder spasm (Renal and urinary disorders) | 1 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Micturition urgency (Renal and urinary disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 1 | 1
Hypertension (Vascular disorders) | 1 | 2
Hypotension (Vascular disorders) | 1 | 0
Venous stasis (Vascular disorders) | 1 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 2
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 0
Device breakage (Injury, poisoning and procedural complications) | 1 | 0
Excoriation (Injury, poisoning and procedural complications) | 1 | 0
Radiation injury (Injury, poisoning and procedural complications) | 1 | 1
Blood bilirubin increased (Investigations) | 1 | 0
Blood creatinine increased (Investigations) | 1 | 0
Blood glucose increased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 1 | 1
Blood urea increased (Investigations) | 1 | 0
International normalised ratio increased (Investigations) | 1 | 0
Prothrombin time prolonged (Investigations) | 1 | 0
Amenorrhoea (Reproductive system and breast disorders) | 1/69 | 0
Epididymitis (Reproductive system and breast disorders) | 1/61 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1/69 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Vertigo (Ear and labyrinth disorders) | 1 | 0
Tachycardia (Cardiac disorders) | 1 | 1
Dry eye (Eye disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2
Aphthous stomatitis (Gastrointestinal disorders) | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 1
Lip disorder (Gastrointestinal disorders) | 0 | 1
Oral mucosal discolouration (Gastrointestinal disorders) | 0 | 1
Salivary gland enlargement (Gastrointestinal disorders) | 0 | 1
Chills (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Mass (General disorders) | 0 | 1
Candidiasis (Infections and infestations) | 0 | 1
Extradural abscess (Infections and infestations) | 0 | 1
Fungal infection (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 1
Oral viral infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 0 | 1
Neuralgia (Nervous system disorders) | 0 | 1
Paraplegia (Nervous system disorders) | 0 | 1
Spinal cord disorder (Nervous system disorders) | 0 | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 0 | 1
Stasis dermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Pharyngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Flushing (Vascular disorders) | 0 | 2
Breath sounds abnormal (Investigations) | 0 | 1
Electrocardiogram Qrs complex abnormal (Investigations) | 0 | 1
Weight decreased (Investigations) | 0 | 1
Weight increased (Investigations) | 0 | 1
Euphoric mood (Psychiatric disorders) | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 1
Pancytopenia (Blood and lymphatic system disorders) | 0 | 1
Neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Polycythaemia vera (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Right ventricular hypertrophy (Cardiac disorders) | 0 | 1
Sinus tachycardia (Cardiac disorders) | 0 | 1
Radiation mucositis (Injury, poisoning and procedural complications) | 0 | 1
Glucose tolerance impaired (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1
Renal impairment (Renal and urinary disorders) | 0 | 1
Urinary incontinence (Renal and urinary disorders) | 0 | 1
Vaginal ulceration (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No